CLINICAL TRIAL: NCT06027970
Title: Efficacy of Continuous Terlipressin Therapy After Endoscopic Variceal Ligation in Acute Variceal Haemorrhage: A Randomised Control Clinical Trial
Brief Title: Efficacy of Continuous Terlipressin Therapy After Endoscopic Variceal Ligation
Acronym: TERLEVL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IEC-INT/2023/Study-865
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Variceal Hemorrhage
MeSH Terms: interventions — Terlipressin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): After successful Endoscopic variceal ligation (EVL) the treatment group will receive injection Terlipressin (1 mg IV bolus q 4 hourly) for 2 days. Both the group will receive standard care of therapy.
  Interventions: Drug: Terlipressin
- Control (Placebo Comparator): After successful Endoscopic variceal ligation (EVL) the control group will receive 10 ml of 0.9% normal saline (NS) IV bolus q 4 hourly instead of Terlipressin for 2 days. Both the group will receive standard care of therapy.
  Interventions: Other: 0.9% normal saline (NS)

INTERVENTIONS:
Drug: Terlipressin — After successful Endoscopic variceal ligation (EVL) The treatment group will receive injection Terlipressin (1 mg IV bolus q 4 hourly) for 2 days
  Other Names: Standard care of therapy; Endoscopic variceal ligation (EVL)
  Arms: Treatment
Other: 0.9% normal saline (NS) — After successful Endoscopic variceal ligation (EVL) the control group will receive 10 ml of 0.9% normal saline (NS) IV bolus q 4 hourly instead of Terlipressin for 2 days
  Arms: Control

SUMMARY:
Upper gastrointestinal (UGI) bleed of variceal origin is a common medical emergency. Prompt endoscopic variceal ligation (EVL) is therapeutic as well as diagnostic. Terlipressin, a vasopressin analog (intravenous, 2 mg q 4 hourly), is widely used promptly in any suspicious cases of variceal haemorrhage (VH) before endoscopic intervention, along with volume and blood resuscitative measures.

As per guideline, after EVL Terlipressin therapy (1 mg IV q 4 hourly) is advised to continue for 2-5 day to prevent re-bleed and mortality [1]. But the prolong use of Terlipressin is not completely safe as well as it is expensive also in resource constraint setting. At present, no randomized control clinical trial (RCT) is available to prove the efficacy of post-EVL Terlipressin therapy in preventing re-bleed and mortality in acute variceal haemorrhage.

During the post marketing surveillance Terlipressin therapy was found to be associated with life threatening complication like cardiac arrhythmia, myocardial ischemia, critical vasoconstriction of peripheral as well as internal organ leading to ischemia or gangrene, severe hyponatremia, hypertension, fluid overload and pulmonary oedema (2-4).

So the justification of continuing Terlipressin for 5 days after EVL is questionable, as the haemostasis is primarily achieved by EVL and the risk versus benefit of Trelipressin therapy after EVL is still unknown. Continue IV Terlipressin therapy also prolongs in-hospital care causing further increase of health care burden.

As per recently concluded institutional study, continuing Terlipressin after EVL in acute VH did not prevent re-bleed or mortality, rather it increased the risk of ADR, duration of hospital stay, in-hospital complications and cost of the therapy [5]. But the study was open level with relatively smaller sample size.

There is still lack of RCT on post-EVL Terlipressin therapy, regarding its efficacy in preventing re-bleed and mortality. So, we have planned this study to evaluate the efficacy of continuous Terlipressin therapy after EVL, in acute VH.

It will be a double blind randomized controlled clinical trial. The study will be carried out in the 2 arms; denoting the duration of Terlipressin therapy after EVL. Participant with acute VH will be randomized into two study groups after successful EVL.

The treatment group will receive injection Terlipressin (1 mg IV bolus q 4 hourly) for 2 days and the control group will receive 10 ml of 0.9% normal saline (NS) IV bolus q 4 hourly instead of Terlipressin for 2 days. Both the group will receive standard care of therapy and will be followed up for 8 weeks. The participants and the recruiter/PI will be unaware of intervention (terlipressin or NS) receiving.

The study will enlighten us regarding efficacy of continuous Terlipressin therapy after EVL to prevent re- bleed and mortality in acute VH. The study will also generate significant data regarding adverse drug events (ADE) and cost effectiveness or pharmaco- economics of continue Terlipressin therapy after EVL.

In the Indian population there is no study to determine the role gene related to variceal bleed or re-bleed. Endothelial dysfunction is the major contributor for the development of portal hypertension and subsequent varices formation in patient with cirrhosis. Development of blood vessel and endothelial function, endothelial proliferation and neoangiogenesis are regulated by vascular endothelial growth factor (VEGF) family genes. In a recently published study, VEGF C(+405)G(rs2010963) single nucleotide polymorphism (SNP) genotype was found to be associated with higher risk of esophageal and gastric varices and bleeding [10]. Since VEGF is the major factor to endothelial proliferation and neoangiogenesis. So, in this study, as a secondary objective, we will also try to explore the association of VEGF genotype with variceal bleed/ re-bleed and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Irrespective of gender
* age ≥ 18 years
* all the patients with endoscopy proven acute VH with successful EVL done

Exclusion Criteria:

* Patients not receiving pre-EVL Terlipressin therapy
* not achieving haemostasis during EVL
* EVL done beyond 48 hours of admission because of hemodynamic instability or encephalopathy
* Patients with chronic kidney disease
* Patients with pregnancy
* Patients who are receiving blood thinners like anti-platelets, anti-coagulation agents within 4 weeks of presentation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Re-bleed | 7 days
  Re-bleed is defined as any significant UGI haemorrhage after EVL, leading to repeat endoscopy, haemodynamic instability and significant drop of haemoglobin requiring blood transfusion.
Mortality | 7 days
  Incidence of episode of mortality

SECONDARY OUTCOMES:
Duration of hospital stay | 1 week
  Number of days of stay in the hospital
need for blood transfusions | 1 week
  After successful EVL, requirement of blood transfusion
Adverse drug reaction (ADR) | 1 week
  Incidence of adverse drug reaction (ADR)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Post Graduate Institute of Medical Education and Research,, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No